CLINICAL TRIAL: NCT03101462
Title: A Randomized, Open-Label, Study to Evaluate the Immunogenicity of One Dose of Live Attenuated Influenza Vaccine (LAIV) Compared to One Dose of Trivalent Inactivated Influenza Vaccine (IIV) in Adults 18-49 Years of Age
Brief Title: Live Attenuated Influenza Vaccine (LAIV) Versus Trivalent Inactivated Influenza Vaccine in Healthy Adults 18-49 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Principal Investigator, Daniel Hoft, MD, PhD, Director, Division of Infectious Diseases, Allergy & Immunology, St. Louis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16354
Record Dates: First submitted 2017-03-23; First posted 2017-04-05 (Actual); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2018-11

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of two different groups to receive either licensed inactivated influenza vaccine (IIV) or licensed live attenuated influenza vaccine (LAIV) from the 2010-2011 season.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): One dose of 0.5 mL Licensed Inactivated Influenza Vaccine (IIV) on Day 0
  Interventions: Biological: Inactivated Influenza Vaccine
- Group 2 (Active Comparator): One dose of 0.5 mL Licensed Live Attenuated Influenza Vaccine (LAIV) on Day 0
  Interventions: Biological: Live Attenuated Influenza Vaccine

INTERVENTIONS:
Biological: Inactivated Influenza Vaccine
  Other Names: IIV
  Arms: Group 1
Biological: Live Attenuated Influenza Vaccine
  Other Names: LAIV
  Arms: Group 2

SUMMARY:
This randomized, open-label, single-site study at Saint Louis University will enroll approximately 40 subjects who are healthy, 18 to 49 years old. Subjects will be randomized in a 1:1 fashion to receive either licensed trivalent FluMist containing (2010-2011 season appropriate), or licensed inactivated trivalent influenza vaccine (2010-2011 season appropriate) so that approximately 20 subjects will be randomized to receive LAIV, and 20 will receive IIV.

DETAILED DESCRIPTION:
This Phase IV, randomized, open-label, single-site study at Saint Louis University will enroll approximately 40 subjects who are healthy, 18 to 49 years old. Subjects will be randomized in a 1:1 fashion to receive either licensed inactivated influenza vaccine (IIV) (2010-2011 season appropriate) or licensed live attenuated influenza vaccine (LAIV) (2010-2011 season appropriate) so that approximately 20 subjects will be randomized to receive IIV, and 20 will receive LAIV. Subjects will receive 1 dose of IIV or LAIV in the Center for Vaccine Development on Day 0 and will return to the site on days 7 and 45 to assess immunogenicity. Subjects will be asked to report any serious adverse events. Blood samples and nasal washes for assessment of immune responses will be obtained at three time points: on Day 0 prior to dosing with IIV or LAIV, and at visits conducted 7 and 45-51 days post vaccination. The study will be conducted just prior to and during the influenza season. Subjects will receive a single dose of IIV or LAIV administered as instructed per package insert. Two contacts will be made with subjects, either telephone calls or e-mail, to collect serious adverse events only, one at Days 28-35, and one at approximately Days 180-190 to conclude the subject's participation. The duration of each subject's participation is approximately 6 months. The primary immune studies conducted with collected samples will include serum hemagglutinin inhibition (HAI) antibody titers, nasal wash influenza-specific secretory immunoglobulin A (IgA) responses, peripheral blood interferon gamma (IFN-γ) ELISPOT assays and peripheral blood carboxyfluorescein succinimidyl ester (CFSE) dilution/intracellular cytokine staining flow cytometric assays. In addition, frozen serum and peripheral blood mononuclear cells (PBMC) samples will be used in exploratory assays to determine the kinetics and nature of innate responses and the detailed molecular signatures of memory T cells induced by IIV and LAIV vaccinations. Investigators will be performing genome-wide expression studies, but will not perform DNA sequencing and will not send anything other than coded samples outside of Saint Louis University.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 to 49 years, inclusive, on the day of randomization (reached his or her 18th year birthday but not yet reached his or her 50th year birthday) at the time of the dose of study product
* Written informed consent and a locally required authorization (eg, HIPAA in the USA, ) obtained from the subject prior to performing any protocol-related procedures.
* Females of child-bearing potential, (ie, unless surgically sterile [eg, bilateral tubal ligation, bilateral oophorectomy, or hysterectomy], has sterile male partner, is at least 1 year post-menopausal, or practices abstinence) must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, or use of a condom with spermicide by the sexual partner) for 30 days prior to the first dose of study product, and must agree to continue using such precautions for 60 days after the dose of vaccine due to a potential dose of live vaccine product. In addition, the subject must also have a negative urine or blood pregnancy test at screening and, if screening and Day 0 do not occur on the same day, a negative urine pregnancy test on the day of vaccination prior to randomization. Investigator judgment is required to assess a female subject's capability of pregnancy.
* Are in good health, as determined by vital signs, medical history to ensure any existing medical diagnoses or conditions are stable and not considered clinically significant by physician investigator, and targeted physical examination based on medical history.
* Able to complete follow-up period of 180 days post dose of vaccine as required by the protocol
* Subject available by telephone
* Able to understand and comply with the requirements of the protocol, as judged by the investigator

Exclusion Criteria:

Any of the following would exclude the subject from participation in the study:

* Have an acute illness, including an oral temperature ≥ 100.4°F, within 3 days prior to vaccination.
* Participated in an investigational influenza vaccine study or had a known infection with "flu" since 2007 (confirmed by laboratory culture, including subtype of the influenza A virus (H1N1) investigational vaccines or illness).
* Previous vaccination against influenza in 2007, 2008, 2009 or 2010 with seasonal trivalent live or inactivated influenza vaccine (including H1N1 vaccines).
* Current or expected receipt of immunosuppressive medications (inhaled and topical corticosteroids are permitted) including corticosteroids (≥ 20 mg/day of prednisone equivalent given daily or on alternate days for ≥ 14 days) within a 30 day window around dose of study vaccine product Note: topical corticosteroids for uncomplicated dermatitis may be used throughout the study according to the judgment of the investigator; topical calcineurin inhibitors may be used in accordance with their package insert at entry and during study participation.
* Receipt of immunoglobulin or blood products within 90 days before randomization into the study or expected receipt during study participation
* Received an experimental agent within 1 month prior to vaccination in this study or expect to receive an experimental agent during the active study period (prior to Day 60 after vaccination (Experimental agent includes: vaccine, biologic, device, or medication).
* Have received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 60 days following the vaccination.
* Any known immunosuppressive condition or immune deficiency disease including known cancer illness or organ transplant
* Have known active HIV, Hepatitis B or Hepatitis C infection.
* Have a known allergy to eggs or other components of the vaccine (including gelatin, formaldehyde, octoxinol, thimerosal, gentamycin and chicken protein) or severe reactions to previous influenza vaccinations.
* History of Guillain-Barré syndrome
* Use of antiviral agents with activity against influenza virus (including amantadine, rimantadine, oseltamivir and zanamivir) within 30 days prior to dose of study vaccine products or anticipated use within 30 days after vaccination
* Breastfeeding woman
* History of alcohol or drug abuse that, in the opinion of the investigator, would affect the subject's safety or compliance with study
* Previous medical history, evidence of an intercurrent illness or any condition that, in the opinion of the investigator, would interfere with evaluation of the study vaccine products or interpretation of subject safety or that may compromise the safety of the subject in the study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2011-02-24 (Actual); Primary Completion 2011-05-13 (Actual); Study Completion 2011-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Hoft, MD, PhD, Principal Investigator — St. Louis University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoft DF, Lottenbach KR, Blazevic A, Turan A, Blevins TP, Pacatte TP, Yu Y, Mitchell MC, Hoft SG, Belshe RB. Comparisons of the Humoral and Cellular Immune Responses Induced by Live Attenuated Influenza Vaccine and Inactivated Influenza Vaccine in Adults. Clin Vaccine Immunol. 2017 Jan 5;24(1):e00414-16. doi: 10.1128/CVI.00414-16. Print 2017 Jan. PMID 27847366

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1 Inactivated Influenza Vaccine (IIV): Subjects aged 18-49 years received one dose of Inactivated Influenza Vaccine (IIV) intramuscularly.
- Group 2 Live Attenuated Influenza Vaccine (LAIV): Subjects 18-49 years of age received one dose of Live Attenuated Influenza Vaccine (LAIV) intranasally.
Period: Overall Study
Arm/Group | Group 1 Inactivated Influenza Vaccine (IIV) | Group 2 Live Attenuated Influenza Vaccine (LAIV)
Started | 19 | 19
Completed | 18 | 18
Not Completed | 1 | 1
Not completed — Missed Visit 02 and/or Visit 03 | 1 | 1

BASELINE CHARACTERISTICS:
Population: In the IIV group, 18 subjects completed Visit 02 and 18 subjects completed Visit 03.
  In the LAIV group, 18 subjects completed Visit 02 and 18 subjects completed Visit 03.
Groups:
- Inactivated Influenza Vaccine (IIV): Eighteen subjects received one dose 0.5 mL of Inactivated Influenza Vaccine intramuscularly on Day 0.
- Live Attenuated Influenza Vaccine (IIV): Eighteen subjects received one dose 0.5 mL Live Attenuated Influenza Vaccine intranasally on Day 0.
- Total: Total of all reporting groups
Arm/Group | Inactivated Influenza Vaccine (IIV) | Live Attenuated Influenza Vaccine (IIV) | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 8 | 10 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 17 | 19 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 4 | 13
  White | 9 | 14 | 23
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Age [Mean (Standard Deviation); unit: years] | 33.5 (10.8) | 30.4 (9.8) | 31.2 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Serum Antibody Responses
Description: Geometric mean hemagglutination inhibition titers to three different influenza viruses
Time Frame: Day 0, Day 7, and Day 45
Population: For IIV group, 18 subjects completed Visit 02 and 18 subjects completed Visit 03.
  For LAIV group, 18 subjects completed Visit 02 and 18 subjects completed Visit 03
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- Inactivated Influenza Vaccine (IIV): One 0.5 mL dose of IIV given intramuscularly.
- Live Attenuated Influenza Vaccine (LAIV): One 0.5 mL dose of LAIV given intranasally.
Arm/Group | Inactivated Influenza Vaccine (IIV) | Live Attenuated Influenza Vaccine (LAIV)
Number analyzed (Participants) | 19 | 19
Titers
  Influenza A virus subtype H1N1 (A/H1N1) Day 0 | 11.76 [6.2 to 22.4] | 11.11 [6.3 to 19.9]
  A/H1N1 Day 7: number analyzed (Participants) | 18 | 18
  A/H1N1 Day 7 | 47.03 [24.3 to 91.1] | 9.33 [5.4 to 16.3]
  A/H1N1 Day 45: number analyzed (Participants) | 18 | 18
  A/H1N1 Day 45 | 101.59 [51.6 to 200] | 12.70 [7.0 to 23.2]
  Influenza A virus subtype H3N2 (A/H3N2) Day 0 | 6.35 [4.1 to 9.9] | 7.44 [4.6 to 12.0]
  A/H3N2 Day 7: number analyzed (Participants) | 18 | 18
  A/H3N2 Day 7 | 17.96 [10.5 to 30.8] | 7.13 [4.1 to 11.7]
  A/H3N2 Day 45: number analyzed (Participants) | 18 | 18
  A/H3N2 Day 45 | 32.00 [17.5 to 58.4] | 9.70 [5.9 to 16.0]
  Influenza B Day 0 | 7.41 [5.2 to 10.6] | 10.71 [6.6 to 17.5]
  Influenza B Day 7: number analyzed (Participants) | 18 | 18
  Influenza B Day 7 | 21.77 [14.2 to 33.4] | 11.31 [6.8 to 18.77]
  Influenza B Day 45: number analyzed (Participants) | 18 | 18
  Influenza B Day 45 | 40.32 [24.4 to 66.7] | 12.70 [7.9 to 20.5]
Statistical Analysis 1: Comparison: Inactivated Influenza Vaccine (IIV) vs Live Attenuated Influenza Vaccine (LAIV); A/H1N1 Day 0; Test type: Other — ANOVA; p = 0.89, t-test, 2 sided
Statistical Analysis 2: Comparison: Inactivated Influenza Vaccine (IIV) vs Live Attenuated Influenza Vaccine (LAIV); A/H1N1 Day 7; Test type: Other; p = 0.00082, t-test, 2 sided — This is the calculated p-value
Statistical Analysis 3: Comparison: Inactivated Influenza Vaccine (IIV) vs Live Attenuated Influenza Vaccine (LAIV); A/H1N1 Day 45; Test type: Other; p = 0.000076, t-test, 2 sided — This is the calculated p-value
Statistical Analysis 4: Comparison: Inactivated Influenza Vaccine (IIV) vs Live Attenuated Influenza Vaccine (LAIV); A/H3N2 Day 0; Test type: Other; p = 0.63, t-test, 2 sided
Statistical Analysis 5: Comparison: Inactivated Influenza Vaccine (IIV) vs Live Attenuated Influenza Vaccine (LAIV); A/H3N2 Day 7; Test type: Other; p = 0.0186, t-test, 2 sided — This is the calculated p-value
Statistical Analysis 6: Comparison: Inactivated Influenza Vaccine (IIV) vs Live Attenuated Influenza Vaccine (LAIV); A/H3N2 Day 45; Test type: Other; p = 0.0052, t-test, 2 sided — This is the calculated p-value
Statistical Analysis 7: Comparison: Inactivated Influenza Vaccine (IIV) vs Live Attenuated Influenza Vaccine (LAIV); Influenza B Day 0; Test type: Other; p = 0.25, t-test, 2 sided
Statistical Analysis 8: Comparison: Inactivated Influenza Vaccine (IIV) vs Live Attenuated Influenza Vaccine (LAIV); Influenza B Day 7; Test type: Other; p = 0.061, t-test, 2 sided
Statistical Analysis 9: Comparison: Inactivated Influenza Vaccine (IIV) vs Live Attenuated Influenza Vaccine (LAIV); Influenza B Day 45; Test type: Other; p = 0.0025, t-test, 2 sided

2. Primary Outcome: T-cell Responses
Description: Number of Interferon gamma ELISPOT spot forming cells (SFC) per million Peripheral Blood Mononuclear Cells (PBMCs) were calculated.
Time Frame: Day 0, Day 7, and Day 45
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Cells/Million PBMC
Arm/Group | Inactivated Influenza Vaccine (IIV) | Live Attenuated Influenza Vaccine (LAIV)
Number analyzed (Participants) | 19 | 19
Cells/Million PBMC
  Medium Alone Day 0 | 1.53 (0.51) | 2.51 (1.05)
  Medium Alone Day 7: number analyzed (Participants) | 18 | 18
  Medium Alone Day 7 | 6.17 (4.21) | 1.05 (0.29)
  Medium Alone Day 45: number analyzed (Participants) | 18 | 18
  Medium Alone Day 45 | 1.11 (0.31) | 2.35 (0.90)
  Peptide Pool 1 + Peptide Pool 2 Day 0 | 75.55 (23.12) | 61.52 (17.09)
  Peptide Pool 1 + Peptide Pool 2 Day 7: number analyzed (Participants) | 18 | 18
  Peptide Pool 1 + Peptide Pool 2 Day 7 | 88.76 (26.98) | 81.11 (14.55)
  Peptide Pool 1 + Peptide Pool 2 Day 45: number analyzed (Participants) | 18 | 18
  Peptide Pool 1 + Peptide Pool 2 Day 45 | 69.94 (19.03) | 65.55 (15.14)
  Live H3N2 Day 0 | 157.90 (29.93) | 126.20 (28.71)
  Live H3N2 Day 7: number analyzed (Participants) | 18 | 18
  Live H3N2 Day 7 | 256.79 (60.12) | 254.26 (49.36)
  Live H3N2 Day 45: number analyzed (Participants) | 18 | 18
  Live H3N2 Day 45 | 180.99 (35.49) | 146.99 (19.72)
  FluMist Day 0 | 39.26 (12.61) | 43.16 (12.46)
  FluMist Day 7: number analyzed (Participants) | 18 | 18
  FluMist Day 7 | 90.25 (24.83) | 104.81 (43.29)
  Flu Mist Day 45: number analyzed (Participants) | 18 | 18
  Flu Mist Day 45 | 70.00 (21.07) | 49.48 (13.68)
Statistical Analysis 1: Comparison: Inactivated Influenza Vaccine (IIV); Peptide Pool 1 and 2, Day 0 and Day 7; Test type: Other; p = 0.24, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Inactivated Influenza Vaccine (IIV); Peptide Pool 1 and 2, Day 0 and Day 45; Test type: Other; p = 0.76, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Inactivated Influenza Vaccine (IIV); Live H3N2, Day 0 and Day 7; Test type: Other; p = 0.06, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Inactivated Influenza Vaccine (IIV); Live H3N2, Day 0 and Day 45; Test type: Other; p = 0.56, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Inactivated Influenza Vaccine (IIV); Flumist, Day 0 and Day 7; Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Inactivated Influenza Vaccine (IIV); Flumist, Day 0 and Day 45; Test type: Other; p = 0.16, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Live Attenuated Influenza Vaccine (LAIV); Peptide Pool 1 and 2, Day 0 and Day 7; Test type: Other; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Live Attenuated Influenza Vaccine (LAIV); Peptide Pool 1 and 2, Day 0 and Day 45; Test type: Other; p = 0.94, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Live Attenuated Influenza Vaccine (LAIV); Live H3N2, Day 0 and Day 7; Test type: Other; p = 0.002, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Live Attenuated Influenza Vaccine (LAIV); Live H3N2, Day 0 and Day 45; Test type: Other; p = 0.16, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Live Attenuated Influenza Vaccine (LAIV); Flumist, Day 0 and Day 7; Test type: Other; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Live Attenuated Influenza Vaccine (LAIV); Flumist, Day 0 and Day 45; Test type: Other; p = 0.98, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Cluster of Differentiation 4 (CD4+) T Cells That Proliferate and Produce Interferon (IFN)-Gamma After Antigen Activation
Description: Mean absolute numbers of CD4(+), Carboxyfluorescein succinimidyl ester [CFSE(low)] IFN-gamma(+), and T cells after activation with a specific antigen measured by flow cytometry
Time Frame: Day 0, Day 7, and Day 45
Population: as for outcome 1
Measure: Mean (Standard Error); unit: T Cells
Arm/Group | Inactivated Influenza Vaccine (IIV) | Live Attenuated Influenza Vaccine (LAIV)
Number analyzed (Participants) | 19 | 19
T Cells
  Medium Day 0 | 92.79 (38.19) | 83.80 (20.60)
  Medium Day 7: number analyzed (Participants) | 18 | 18
  Medium Day 7 | 1075.24 (711.71) | 65.45 (18.04)
  Medium Day 45: number analyzed (Participants) | 18 | 18
  Medium Day 45 | 338.86 (224.16) | 144.58 (64.94)
  Live H3N2 Day 0 | 15939.07 (5984.03) | 22958.77 (8371.46)
  Live H3N2 Day 7: number analyzed (Participants) | 18 | 18
  Live H3N2 Day 7 | 32527.86 (11165.21) | 28557.23 (8835.01)
  Live H3N2 Day 45: number analyzed (Participants) | 18 | 18
  Live H3N2 Day 45 | 21320.85 (6054.77) | 15654.57 (4626.64)
  FluMist Day 0 | 14009.94 (6259.10) | 12552.22 (3718.47)
  Flu Mist Day 7: number analyzed (Participants) | 18 | 18
  Flu Mist Day 7 | 26999.98 (9510.82) | 24265.06 (5147.71)
  Flu Mist Day 45: number analyzed (Participants) | 18 | 18
  Flu Mist Day 45 | 21704.19 (6455.24) | 14618.15 (4314.62)
Statistical Analysis 1: Comparison: Inactivated Influenza Vaccine (IIV); Peptide Pool 1 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 7; Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Inactivated Influenza Vaccine (IIV); Peptide Pool 1 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 45; Test type: Other; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Inactivated Influenza Vaccine (IIV); Peptide Pool 2 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 7; Test type: Other; p = 0.95, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Inactivated Influenza Vaccine (IIV); Peptide Pool 2 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 45; Test type: Other; p = 0.17, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Inactivated Influenza Vaccine (IIV); Peptide Pool 1 and Peptide Pool 2 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 7; Test type: Other; p = 0.06, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Inactivated Influenza Vaccine (IIV); Peptide Pool 1 and Peptide Pool 2 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 45; Test type: Other; p = 0.14, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Inactivated Influenza Vaccine (IIV); Live H3N2 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 7; Test type: Other; p = 0.02, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Inactivated Influenza Vaccine (IIV); Live H3N2 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 45; Test type: Other; p = 0.09, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Inactivated Influenza Vaccine (IIV); Flumist CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 7; Test type: Other; p = 0.01, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Inactivated Influenza Vaccine (IIV); Flumist CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 45; Test type: Other; p = 0.08, Wilcoxon (Mann-Whitney)
Statistical Analysis 11: Comparison: Live Attenuated Influenza Vaccine (LAIV); Peptide Pool 1 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 7; Test type: Other; p = 0.16, Wilcoxon (Mann-Whitney)
Statistical Analysis 12: Comparison: Live Attenuated Influenza Vaccine (LAIV); Peptide Pool 1 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 45; Test type: Other; p = 0.76, Wilcoxon (Mann-Whitney)
Statistical Analysis 13: Comparison: Live Attenuated Influenza Vaccine (LAIV); Peptide Pool 2 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 7; Test type: Other; p = 0.84, Wilcoxon (Mann-Whitney)
Statistical Analysis 14: Comparison: Live Attenuated Influenza Vaccine (LAIV); Peptide Pool 2 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 45; Test type: Other; p = 0.04, Wilcoxon (Mann-Whitney)
Statistical Analysis 15: Comparison: Live Attenuated Influenza Vaccine (LAIV); Peptide Pool 1 and Peptide Pool 2 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 7; Test type: Other; p = 0.07, Wilcoxon (Mann-Whitney)
Statistical Analysis 16: Comparison: Live Attenuated Influenza Vaccine (LAIV); Peptide Pool 1 and Peptide Pool 2 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 45; Test type: Other; p = 0.27, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: Live Attenuated Influenza Vaccine (LAIV); Live H3N2 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 7; Test type: Other; p = 0.11, Wilcoxon (Mann-Whitney)
Statistical Analysis 18: Comparison: Live Attenuated Influenza Vaccine (LAIV); Live H3N2 CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 45; Test type: Other; p = 0.46, Wilcoxon (Mann-Whitney)
Statistical Analysis 19: Comparison: Live Attenuated Influenza Vaccine (LAIV); Flumist CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 7; Test type: Other; p = 0.006, Wilcoxon (Mann-Whitney)
Statistical Analysis 20: Comparison: Live Attenuated Influenza Vaccine (LAIV); Flumist CD4+/CFSE(low)/IFN-gamma+, Day 0 and Day 45; Test type: Other; p = 0.41, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Secretory Immunoglobulin A (IgA) Responses
Description: Influenza virus strain-specific nasal wash secretory immunoglobulin A (IgA) titers by ELISA was measured
Time Frame: Day 0 and Day 45
Population: For IIV group, 18 subjects completed Visit 03. For LAIV group, 18 subjects completed Visit 03.
Measure: Median (95% Confidence Interval); unit: Titers
Arm/Group | Inactivated Influenza Vaccine (IIV) | Live Attenuated Influenza Vaccine (LAIV)
Number analyzed (Participants) | 19 | 19
Titers
  Influenza A/H1N1 Day 0 | 18 [1.25 to 64] | 16.25 [3 to 41]
  Influenza A/H1N1 Day 45: number analyzed (Participants) | 18 | 18
  Influenza A/H1N1 Day 45 | 20.75 [1.25 to 2328] | 28.5 [4 to 197]
  Influenza A/H3N2 Day 0 | 26.5 [5 to 69] | 32.25 [1.25 to 88]
  Influenza A/H3N2 Day 45: number analyzed (Participants) | 18 | 18
  Influenza A/H3N2 Day 45 | 31.5 [3 to 476] | 57.25 [10 to 458]
  Influenza B Day 0 | 16 [3 to 50] | 9.75 [3 to 47]
  Influenza B Day 45: number analyzed (Participants) | 18 | 18
  Influenza B Day 45 | 16.5 [1.25 to 77] | 16.75 [5 to 113]
Statistical Analysis 1: Comparison: Inactivated Influenza Vaccine (IIV); Influenza A/H1N1 HA, Day 0 and Day 45; Test type: Other; p = 0.72, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Inactivated Influenza Vaccine (IIV); Influenza A/H3N2 HA, Day 0 and 45; Test type: Other; p = 0.06, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Inactivated Influenza Vaccine (IIV); Influenza B HA, Day 0 and Day 45; Test type: Other; p = 0.75, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Live Attenuated Influenza Vaccine (LAIV); Influenza A/H1N1 HA, Day 0 and Day 45; Test type: Other; p = 0.05, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Live Attenuated Influenza Vaccine (LAIV); Influenza A/H3N2 HA, Day 0 and Day 45; Test type: Other; p = 0.0004, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Live Attenuated Influenza Vaccine (LAIV); Influenza B HA, Day 0 and Day 45; Test type: Other; p = 0.02, Wilcoxon (Mann-Whitney)

5. Primary Outcome: Hemagglutinin Immunoglobulin A (IgA) Responses
Description: Hemagglutinin (HA) specific nasal wash secretory immunoglobulin A (IgA) of serum reactivity with HA bound to ELISA plates.
Time Frame: Day 7
Measure: Mean (Standard Error); unit: Fold change
Arm/Group | Inactivated Influenza Vaccine (IIV) | Live Attenuated Influenza Vaccine (LAIV)
Number analyzed (Participants) | 18 | 18
Fold change
  IgA anti-H1N1 HA Day 7 | 2.32 (0.40) | 8.42 (3.51)
  IgA anti-H3N2 Day 7 | 1.77 (0.24) | 9.42 (4.98)
  IgA anti-Influenza B Day 7 | 1.94 (0.58) | 9.55 (4.52)
Statistical Analysis 1: Comparison: Inactivated Influenza Vaccine (IIV) vs Live Attenuated Influenza Vaccine (LAIV); Fold increase IgA anti-H1N1 HA, Day 7; Test type: Other; p = 0.02, Fisher Exact
Statistical Analysis 2: Comparison: Inactivated Influenza Vaccine (IIV) vs Live Attenuated Influenza Vaccine (LAIV); Fold increase IgA anti-H3N2, Day 7; Test type: Other; p = 0.67, Fisher Exact
Statistical Analysis 3: Comparison: Inactivated Influenza Vaccine (IIV) vs Live Attenuated Influenza Vaccine (LAIV); Fold increase IgA anti-influenza B HA, Day 7; Test type: Other; p = 0.30, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Day 0 through Day 28. Serious Adverse Events were collected from Day 0 through Day 180.
Groups:
- Group 1 Licensed Trivalent FluMist: Subjects received one dose of Licensed Trivalent FluMist at Day 0.
- Group 1 Inactvated Trivalent Influenza Vaccine: Subjects received one dose of Inactivated Trivalent Influenza Vaccine at Day 0.
Arm/Group | Group 1 Licensed Trivalent FluMist | Group 1 Inactvated Trivalent Influenza Vaccine
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 1/19 | 0/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 Licensed Trivalent FluMist (N=19) | Group 1 Inactvated Trivalent Influenza Vaccine (N=18)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes